CLINICAL TRIAL: NCT04684420
Title: A Randomized Phase I, Open-Label, Active-Controlled Study Assessing The BE Between Single Doses of 500 mg GXR RM Tablets and 500 mg GXR Tablets Under Fasted and Fed State in Two 2-Way Crossover Groups of Healthy Participants
Brief Title: GXR RM (Glucophage® Extended Release Reduced Mass) 500 Milligram (mg) Korea Bioequivalence (BE) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200084_0028
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Diabetes Mellitus; Glucophage Extended Release; Bioequivalence Study
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Reference GXR (Fasting), Then Test GXR RM (Fasting) (Experimental): Participants received a single oral dose of 500 milligram (mg) of reference GXR (Glucophage® Extended Release) tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg test GXR RM (Reduced Mass) tablet on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
  Interventions: Drug: Glucophage® XR RM Test; Drug: Glucophage® XR Reference
- First Test GXR RM (Fasting), Then Reference GXR (Fasting) (Experimental): Participants received a single oral dose of 500 milligrams (mg) of test GXR RM tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg of reference GXR tablet on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
  Interventions: Drug: Glucophage® XR RM Test; Drug: Glucophage® XR Reference
- First Reference GXR (Fed), Then Test GXR RM (Fed) (Experimental): Participants received a single oral dose of 500 milligrams (mg) of reference GXR tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg of test GXR RM tablet on Day 8 in treatment period 2 under fed conditions. There was a washout period of 7 days between two treatment period.
  Interventions: Drug: Glucophage® XR RM Test; Drug: Glucophage® XR Reference
- First Test GXR RM (Fed), Then Reference GXR (Fed) (Experimental): Participants received a single oral dose of 500 milligrams (mg) of test GXR RM tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg of reference GXR tablet on Day 8 in treatment period 2 under fed conditions. There was a washout period of 7 days between two treatment period.
  Interventions: Drug: Glucophage® XR RM Test; Drug: Glucophage® XR Reference

INTERVENTIONS:
Drug: Glucophage® XR RM Test — Participants received a single oral dose of 500 mg of test Glucophage® XR RM tablet under fasting or fed conditions.
  Other Names: Metformin hydrochloride
Drug: Glucophage® XR Reference — Participants received a single oral dose of 500 mg of reference Glucophage® XR tablet under fasting or fed conditions.
  Other Names: Metformin hydrochloride

SUMMARY:
The purpose of this study was to assess bioequivalence (BE) of newly developed Glucophage® XR (GXR) reduced mass (RM) tablet (metformin hydrochloride 500 milligrams (mg) test tablet) and marketed Glucophage ® XR tablet (metformin hydrochloride 500 mg reference tablet) following single oral dose administration under fasted and fed conditions by comparing pharmacokinetics, safety and tolerability between test and reference in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* All values for hematology and biochemistry tests of blood and urinalysis (especially Estimated Glomerular Filtration Rate [eGFR] greater than [>] 80 milliliters per minute per 1.73 square meter [80 ml/min/1.73 m^2] and normal Creatinine) within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Are not having congenital or chronic diseases, nor pathological symptoms based on the screening
* Have no history of gastrointestinal resection that may affect drug absorption
* Have no history of psychiatric disorder within 5 years prior to screening
* Vital signs (body temperature [tympanic], blood pressure [BP], and pulse rate in sitting position) within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Electrocardiogram recording (12-lead) without signs of clinically relevant pathology in particular QTc (Bazett) less than or equal to [<=] 450 millisecond (ms)
* Non-smoker (that is [i.e.] zero cigarettes, pipes, cigars or others) at least three months before study entry
* Negative screen for Hepatitis B surface antigen (HBsAg) and Hepatitis B Virus antibody (anti-HBc), Hepatitis C Virus antibody (anti-HCV) and Human Immunodeficiency Virus antibodies (anti-HIV 1 and 2) and Rapid Plasma Reagin Antibody (RPR Ab)
* Have a body weight within the range 55 to 95 kilograms (kg) and a Body Mass Index (BMI) within the range 18.5 to 29.9 kilograms per square meter (kg/m^2) (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants determined ineligible to participate in this study at the discretion of the Principal Investigator (or delegated investigators)
* Hypersensitivity to venous puncture
* Known hypersensitivity to ingredients of Study Interventions or Biguanides, or having other clinically relevant hypersensitivities
* Type I diabetes mellitus, lactic acidosis, acute or chronic metabolic acidosis including diabetic ketoacidosis, with or without coma; diabetic pre-coma, pre-diabetes
* Participants with renal impairment (eGFR < 80 ml/min/1.73m^2) - calculations according to Modification of Diet in Renal Disease (MDRD) formula). Participants presenting with acute conditions with the potential to alter renal function such as dehydration, severe infection, cardiovascular collapse (shock), acute myocardial infraction, and septicemia
* Participants with acute and unstable heart failure
* Participants with severe infection or severe traumatic general disorder
* Participants who are scheduled to undergo surgical procedures
* Participants with malnutrition, inanition, pituitary dysfunction or adrenal function failure
* Participants with hepatic dysfunction, acute or chronic disease which may cause tissue hypoxia such as respiratory failure, acute myocardial infarction, shock and gastrointestinal (GI) disorder such as excessive alcohol intake, hydration, diarrhea, vomiting etc.
* Participants undergoing intravascular administration of iodinated contrast materials in radio diagnostic examinations (for example, intravenous urogram, intravenous cholangiography, angiography, and computed tomography (CT) scans with intravascular contrast materials etc.)
* Participants who took drugs that significantly induce (e.g., barbiturate) or inhibit drug metabolism enzymes, and those drugs that may alter metformin pharmacokinetic (pK), most importantly organic cation transporter 1/2 [OCT1/2] inhibitors and inducers, within 30 days prior to screening
* Use of a concomitant drug. However, any medications that are considered necessary for participant's welfare and will not interfere with the trial medication may be given at the discretion of the investigator
* Use of any medication that may affect the outcome of the study within 10 days prior to screening and during study conduct
* Participation in another bioequivalence or other clinical studies where the last administration of previous study medication was within 6 months, before the first drug administration in this study
* Other protocol defined exclusion criteria could apply

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Clinical Trials Center, Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200084_0028
- See also: Medical Information Location Map - Med Info Contact — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 participants were screened for the study in Part 1 (Fasted state) out of which 48 were randomized. For Part 2 (Fed state), a total of 49 participants were screened out of which 33 were randomized.
Groups:
- First Reference GXR (Fasting), Then Test GXR RM Tablet (Fasting): Participants received a single oral dose of 500 milligram (mg) of reference GXR (Glucophage® Extended Release) tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg test GXR RM (Reduced Mass) tablet on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
Period: Treatment Period 1 (Day 1)
Arm/Group | First Reference GXR (Fasting), Then Test GXR RM Tablet (Fasting) | First Test GXR RM (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fed), Then Test GXR RM (Fed) | First Test GXR RM (Fed), Then Reference GXR (Fed)
Started | 24 | 24 | 17 | 16
Completed | 24 | 23 | 15 | 15
Not Completed | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 2(Day 8 up to 3 Months)
Arm/Group | First Reference GXR (Fasting), Then Test GXR RM Tablet (Fasting) | First Test GXR RM (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fed), Then Test GXR RM (Fed) | First Test GXR RM (Fed), Then Reference GXR (Fed)
Started | 24 | 23 | 15 | 15
Completed | 24 | 23 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic population included all those participants who participated in the bioequivalence study (that is all participants who were randomized)
Units Other Than Participants: Count of Participants
Groups:
- First Reference GXR (Fasting), Then Test GXR RM (Fasting): Participants received a single oral dose of 500 mg of reference GXR tablet on Day 1 in treatment period 1 followed by single oral dose of 500 mg test GXR RM tablet on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
- Total: Total of all reporting groups
Arm/Group | First Reference GXR (Fasting), Then Test GXR RM (Fasting) | First Test GXR RM (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fed), Then Test GXR RM (Fed) | First Test GXR RM (Fed), Then Reference GXR (Fed) | Total
Number analyzed (Participants) | 24 | 24 | 17 | 16 | 81
Number analyzed (Count of Participants) | 24 | 24 | 17 | 16 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 17 | 16 | 81
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 5 | 3 | 22
  Male | 17 | 17 | 12 | 13 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 24 | 24 | 17 | 16 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Metformin
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Part 1 (fasted): Pre-dose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24 and 32 hours post dose. Part 2 (fed): Pre-dose 1, 2, 3, 4, 5, 5.5, 6, 6.5, 7, 8, 9, 10, 12, 24 and 32 hours post dose
Population: Pharmacokinetic Analysis Set included those participants who completed investigational medicinal product (IMP) administration and completed all pharmacokinetic blood collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliter (hr*ng/ml)
Groups:
- Reference GXR (Fasting): Participants received a single oral dose of 500 miligrams (mg) of reference GXR tablet either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
- Test GXR RM (Fasting): Participants received a single oral dose of 500 mg of test GXR RM tablet either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
- Reference GXR (Fed): Participants received a single oral dose of 500 mg of reference GXR tablet either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fed conditions. There was a washout period of 7 days between two treatment period.
- Test GXR RM (Fed): Participants received a single oral dose of 500 mg of test GXR RM tablet either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fed conditions. There was a washout period of 7 days between two treatment period.
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 30 | 30
hour*nanogram per milliter (hr*ng/ml) | 3627.171 (31.9) | 4076.521 (30.4) | 6981.833 (18.1) | 6564.938 (26.4)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Reference GXR (Fasting): Participants received a single oral dose of 500 mg of reference GXR tablet either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fasting conditions. There was a washout period of 7 days between two treatment period.
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 30 | 30
nanogram per milliliter (ng/mL) | 605.347 (31.7) | 677.651 (31.2) | 590.956 (18.9) | 671.864 (16.7)

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: From Day 1 up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants
  TEAEs | 7 | 7 | 3 | 2
  Serious TEAEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Taking Concomitant Medications
Description: Concomitant medications included medications administered from the first administration of study interventions to the end of observation.
Time Frame: From Day 1 up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Description: The laboratory measurements included hematology, blood chemistry, urinalysis and Blood Sugar Test (BST). Number of participants with clinically significant changes from baseline in laboratory values were reported. Clinically Significance was decided by investigator.
Time Frame: From Day1 (baseline) up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants
  Hematology | 0 | 0 | 0 | 0
  Biochemistry | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0
  Blood Sugar Test (BST) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported. Clinically significance was decided by investigator.
Time Frame: From Day 1 (baseline) up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate, body temperature and respiration rate. Number of participants with clinically significant changes from baseline in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: From Day 1 (baseline) up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings
Description: Physical examination included assessments of the skin, lungs, cardiovascular system, abdomen (liver and spleen), and the symptoms reported by the participant. Number of participants with clinically significant changes from baseline in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: From Day 1 (baseline) up to 3 weeks
Population: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 48 | 32 | 31
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Metformin
Description: AUC0-inf was calculated by combining AUC0-t and AUC extra. AUC extra represents an extrapolated value obtained by Clast/ lambda z, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and lambda z is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis Set included those participants who completed investigational medicinal product (IMP) administration and completed all pharmacokinetic blood collection. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 29 | 30
hr*ng/ml | 3911.152 (30.8) | 4370.051 (28.6) | 7297.899 (16.4) | 6833.321 (23.6)

10. Secondary Outcome: Ratio of Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-tlast) to Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Metformin
Description: The ratio of AUClast to AUCinf were reported.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 29 | 30
Ratio | 0.927 (4.7) | 0.933 (3.2) | 0.953 (9.9) | 0.961 (3.5)

11. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Metformin
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 29 | 30
hours | 3.520 (60.1) | 3.769 (47.1) | 4.122 (19.5) | 3.386 (21.1)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metformin
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
Number analyzed (Participants) | 47 | 47 | 30 | 30
hours | 3.500 [2.000 to 5.000] | 3.500 [1.000 to 5.000] | 5.500 [4.000 to 10.000] | 5.010 [5.000 to 8.000]

ADVERSE EVENTS:
Time Frame: From informed consent (Day-28 to Day-2) up to 3 weeks, a maximum of 49 days.
Description: The Safety Analysis Set included all participants who administered at least one dose of study interventions.
Arm/Group | Reference GXR (Fasting) | Test GXR RM (Fasting) | Reference GXR (Fed) | Test GXR RM (Fed)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 7/47 | 7/48 | 3/32 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference GXR (Fasting) (N=47) | Test GXR RM (Fasting) (N=48) | Reference GXR (Fed) (N=32) | Test GXR RM (Fed) (N=31)
Human chorionic gonadotropin increased (Investigations) | 2 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 2 | 2 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0
Blood lactic acid increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 3 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04684420/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04684420/SAP_001.pdf